CLINICAL TRIAL: NCT06095505
Title: A Phase 2 Study of Alisertib in Patients With Extensive Stage Small Cell Lung Cancer
Brief Title: A Study of Alisertib in Patients With Extensive Stage Small Cell Lung Cancer
Acronym: ALISCA-Lung1
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Puma Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PUMA-ALI-4201
Record Dates: First submitted 2023-09-27; First posted 2023-10-23 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Small Cell Lung Cancer
Keywords: Alisertib; SCLC
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — MLN 8237

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Alisertib (Experimental): 50 mg (Prior to Amendment 2) or 60 mg (Amendment 2) of alisertib PO BID on days 1-7 of each 21-day cycle
  Interventions: Drug: Alisertib

INTERVENTIONS:
Drug: Alisertib — Alisertib enteric-coated tablets
  Other Names: PB-8237; MLN8237

SUMMARY:
PUMA-ALI-4201 is a Phase 2 study evaluating alisertib monotherapy in patients with pathologically-confirmed small cell lung cancer (SCLC) following progression on or after treatment with one platinum-based chemotherapy and anti-PD-L1 immunotherapy agent. Up to one additional systemic anti-cancer therapy for SCLC is allowed, for a total of up to two prior lines of therapy. This study is intended to identify the biomarker-defined subgroup(s) that may benefit most from alisertib treatment and to evaluate the efficacy, safety, and pharmacokinetics of alisertib.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years at signing of informed consent
* Pathologically confirmed SCLC
* Prior treatment with one platinum-based chemotherapy and an anti-PD-L1 immunotherapy. Up to one additional systemic anti-cancer therapy for SCLC is allowed, for a total of up to two prior lines of therapy

Exclusion Criteria:

* Prior treatment with an AURKA specific-targeted or pan-Aurora-targeted agent, including alisertib in any setting

Note: There are additional inclusion and exclusion criteria. The study center will determine if you meet all of the criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-02-08 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) within biomarker-defined subgroup | From date of first dose to first confirmed Complete or Partial Response, whichever came earlier, assessed up to 36 months
  Objective response rate is defined as the percentage of participants demonstrating a confirmed objective response during the study
Duration of response (DOR) within biomarker-defined subgroup | From start date of response (after date of first dose) to first PD, assessed up to 36 months
  Duration of response is measured from the time at which measurement criteria are first met for CR or PR (whichever status is recorded first) until the first date of recurrence or progressive disease (PD) or death is objectively documented.
Disease Control Rate (DCR) within biomarker-defined subgroup | From date of first dose to first confirmed Complete or Partial Response, whichever came earlier, assessed up to 36 months
  Disease control rate is the proportion of patients who achieve overall tumor response (confirmed CR or PR) or SD lasting for at least 8 weeks from first dose of investigational product.
Progression Free Survival (PFS) within biomarker-defined subgroup | From date of first dose to date of recurrence, progression or death, assessed up to 36 months
  Progression Free Survival (PFS) is measured in months and based on the local tumor assessment. The time interval from the date of first dose until the first date on which recurrence, progression, or death due to any cause, is documented.
Overall Survival (OS) within biomarker-defined subgroup | From date of first dose to death, assessed up to 36 months
  Overall survival (OS) is defined as the time from date of first dose to death due to any cause, censored at the last date known alive on or prior to the data cutoff employed for the analysis, whichever was earlier.

SECONDARY OUTCOMES:
Objective response rate (ORR) in the enrolled patient population | From date of first dose to first confirmed Complete or Partial Response, whichever came earlier, assessed up to 36 months
  Objective response rate is defined as the percentage of participants demonstrating a confirmed objective response during the study.
Duration of response (DOR) in the enrolled patient population | From start date of response (after date of first dose) to first PD, assessed up to 36 months
  Duration of response is measured from the time at which measurement criteria are first met for CR or PR (whichever status is recorded first) until the first date of recurrence or progressive disease (PD) or death is objectively documented.
Disease Control Rate (DCR) in the enrolled patient population | From date of first dose to first confirmed Complete or Partial Response, whichever came earlier, assessed up to 36 months
  Disease control rate is the proportion of patients who achieve overall tumor response (confirmed CR or PR) or SD lasting for at least 8 weeks from first dose of investigational product.
Progression Free Survival (PFS) in the enrolled patient population | From date of first dose to date of recurrence, progression or death, assessed up to 36 months
  Progression Free Survival (PFS) is measured in months and based on the local tumor assessment. The time interval from the date of first dose until the first date on which recurrence, progression, or death due to any cause, is documented.
Overall Survival (OS) in the enrolled patient population | From date of first dose to death, assessed up to 36 months
  Overall survival (OS) is defined as the time from date of first dose to death due to any cause, censored at the last date known alive on or prior to the data cutoff employed for the analysis, whichever was earlier.
Percentage of Participants With Treatment-Emergent Adverse Events (Adverse Events and Serious Adverse Events) in the enrolled patient population | From date of first dose through last dose plus 28 days, assessed up to 36 months
  Treatment emergent adverse events are those events reported on or after the first dose of investigational product and up to 28 days after last dose.

CONTACTS AND LOCATIONS:
Overall Officials: Chief Scientific Officer, Study Director — Puma Biotechnology, Inc.
Locations (30):
- United States (30):
  - Southern Cancer Center, Daphne, Alabama
  - The Oncology Institute of Hope and Innovation, Long Beach, California
  - Rocky Mountain Cancer Centers, Lone Tree, Colorado
  - Georgetown Lombardi Cancer Center, Washington D.C., District of Columbia
  - Clermont Oncology Center, Clermont, Florida
  - The Oncology Institute of Hope and Innovation, Fort Lauderdale, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Illinois Cancer Specialists, Niles, Illinois
  - Indiana University Melvin and Bren Simon Comprehensive Cancer Center, Indianapolis, Indiana
  - University of Maryland Greenebaum Comprehensive Cancer Center, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Minnesota Oncology Hematology, Burnsville, Minnesota
  - Nebraska Cancer Specialists, Grand Island, Nebraska
  - Oncology Hematology Care Clinical Trials, Cincinnati, Ohio
  - University Hospital - Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Zangmeister Cancer Center, Columbus, Ohio
  - Oncology Associates of Oregon, Eugene, Oregon
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina Hollings Cancer Center, Charleston, South Carolina
  - SCRI Oncology Partners, Nashville, Tennessee
  - Texas Oncology-Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Oncology & Hematology Associates of Southwest Virginia, Blacksburg, Virginia
  - Universtity of Virginia Health System, Charlottesville, Virginia
  - Virginia Cancer Specialists Research Institute, Fairfax, Virginia
  - Northwest Cancer Specialists, Vancouver, Washington
  - Marshfield Medical Center, Marshfield, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Puma Biotechnology is committed to sharing clinical trial data and information to help physicians and patients make informed treatment decisions, and to help qualified researchers advance scientific knowledge.
  In accordance with legal and regulatory requirements, Puma publishes study protocol information and clinical study results on clinical trial registries, including ClinicalTrials.gov and EU Clinical Trials Register. Puma also publishes information about clinical studies in peer-reviewed scientific journals and shares data in scientific meetings.
  Puma commits to safeguarding confidentiality and patient privacy throughout the clinical trial data and information sharing process. Any patient-level data will be anonymized to protect personally identifiable information.
  Qualified researchers and study participants may submit requests for other study documentation and clinical trial data to clinicaltrials@pumabiotechnology.com for consideration.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Clinical study documents and clinical trial data may be requested by qualified researchers and study participants for studies that have been completed for at least 18 months, and for which the indication of the drug has been approved in the US and/or EU, as applicable. Requests will be accepted for up to 24 months after the criteria described in this section are met.
Access Criteria: Requestors must provide organizational contact information; a detailed research plan, including outcomes; timeline for completion of the research; qualifications of the research team; funding source; and potential conflicts of interest.
  Puma will not provide access to patient-level data if there is a reasonable likelihood that individual patients could be identified, or in cases where confidentiality or consent provisions prohibit transfer of data or information to third parties. Additionally, Puma will not disclose information that jeopardizes intellectual property rights or divulges confidential commercial information.
URL: https://pumabiotechnology.com/data_sharing_policy.html